CLINICAL TRIAL: NCT00041678
Title: Study of Aripiprazole in the Treatment of Patients With Psychosis Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Purpose: Treatment
Other Study IDs: CN138-005
Record Dates: First submitted 2002-07-12; First posted 2002-07-15 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2007-09

CONDITIONS: Alzheimer Disease
Keywords: Psychosis Associated with Dementia of the Alzheimer's Type
MeSH Terms: conditions — Alzheimer Disease | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The purpose of this study is to learn if aripiprazole is safe and effective in the treatment of psychosis associated with dementia of the Alzheimer's type.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized patients with Alzheimer's Disease

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Local Institution, Rosemead, California
  - Local Institution, Miami, Florida
  - Local Institution, Nashville, Tennessee
  - Local Institution, Bennington, Vermont
  - Local Institution, Burlington, Vermont
  - Local Institution, Milwaukee, Wisconsin